CLINICAL TRIAL: NCT02683928
Title: A Phase IIa, Double-Blind, Randomised, Placebo-controlled, Exploratory Study to Evaluate the Safety, Biological Activity and Pharmacokinetics of GBR 830 in Adults With Moderate-to-Severe Atopic Dermatitis
Brief Title: To Assess the Safety and Activity of GBR 830, Compared to Placebo, in Adults With Moderate-to-severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ichnos Sciences SA (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBR 830-201
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- GBR 830 (Experimental): Two doses of GBR 830, 10 mg/kg (solution for infusion, prepared in normal saline) administered intravenously (IV) four weeks apart.
  Interventions: Biological: GBR 830
- Placebo (Placebo Comparator): Two doses of placebo (formulation buffer for infusion, prepared in normal saline) administered IV four weeks apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBR 830
  Arms: GBR 830
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of GBR 830 on biomarkers in atopic dermatitis to enable further studies in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Atopic dermatitis involvement that of at least 10% body surface area

Exclusion Criteria:

* Treatment with systemic corticosteroids within 4 weeks before randomization, and topical steroids, tacrolimus and/or pimecrolimus within 1 week before the randomization (except emollients, and mild steroids (class 6 or 7)
* Any cell-depleting agents including but not limited to rituximab: within 6 months prior to the baseline visit or until lymphocyte and CD 19+ lymphocyte counts return to normal, whichever is longer. Other biologics: within 5 half-lives or 8 weeks prior to the baseline visit, whichever is longer. Allergen immunotherapy within 6 months before the baseline visit.
* Patient with history of serious local infection and systemic infection Patient with history or current evidence of diseases such as tuberculosis, malignant disease, other inflammatory or autoimmune disease or HIV or Hepatitis B or C positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Wolff, MD, Study Director — Glenmark Pharmaceuticals
Locations (17):
- United States (12):
  - Glenmark Investigational Site 14, Rogers, Arkansas
  - Glenmark Investigational Site 5, Los Angeles, California
  - Glenmark Investigational Site 3, San Diego, California
  - Glenmark Investigational Site 15, Tampa, Florida
  - Glenmark Investigational Site 11, St Louis, Missouri
  - Glenmark Investigational Site 16, Berlin, New Jersey
  - Glenmark Investigational Site 1, New York, New York
  - Glenmark Investigational Site 9, Raleigh, North Carolina
  - Glenmark Investigational Site 13, Fairborn, Ohio
  - Glenmark Investigational Site 2, Dallas, Texas
  - Glenmark Investigational Site 17, Katy, Texas
  - Glenmark Investigational Site 12, Webster, Texas
- Canada (5):
  - Glenmark Investigational Site 8, Markham, Ontario
  - Glenmark Investigational Site 7, Peterborough, Ontario
  - Glenmark Investigational Site 6, Richmond Hill, Ontario
  - Glenmark Investigational Site 10, Waterloo, Ontario
  - Glenmark Investigational Site 4, Montreal, Quebec

REFERENCES:
- [Result] Guttman-Yassky E, Pavel AB, Zhou L, Estrada YD, Zhang N, Xu H, Peng X, Wen HC, Govas P, Gudi G, Ca V, Fang H, Salhi Y, Back J, Reddy V, Bissonnette R, Maari C, Grossman F, Wolff G. GBR 830, an anti-OX40, improves skin gene signatures and clinical scores in patients with atopic dermatitis. J Allergy Clin Immunol. 2019 Aug;144(2):482-493.e7. doi: 10.1016/j.jaci.2018.11.053. Epub 2019 Feb 6. PMID 30738171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GBR 830 | Placebo
Started | 48 | 16
Completed | 26 | 8
Not Completed | 22 | 8

BASELINE CHARACTERISTICS:
Population: A total of 64 eligible participants were randomized to receive either GBR 830 or corresponding placebo. Two participants assigned to GBR 830 withdrew informed consent before dosing. Therefore, a total of 62 subjects were included in the Full Analysis Set and Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | GBR 830 | Placebo | Total
Number analyzed (Participants) | 46 | 16 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (13.38) | 40.4 (15.14) | 37.3 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 5 | 30
  Male | 21 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 42 | 16 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 31 | 11 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.10 (4.086) | 26.23 (3.688) | 26.13 (3.958)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: A treatment-emergent adverse event (TEAE) was defined as any new adverse event (AEs) or worsening of an existing condition after administration of the study drug up to and including the follow-up visit.
Time Frame: 16 weeks
Population: The Safety Analysis Set consisted of all participants who took at least 1 full or partial dose of study treatment and were used in the assessment and reporting of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 46 | 16
Participants
  experiencing at least 1 TEAE | 29 | 10
  experiencing at least 1 SAE | 1 | 0
  TEAE leading to permanent withdrawal of study drug | 2 | 1
  TEAE related to study drug | 4 | 4

2. Primary Outcome: Change From Baseline in Thickness of Lesional Skin Biopsies
Description: Epidermal thickness was assessed in Hematoxylin and Eosin stained sections of lesional skin biopsies on Day 1 (baseline), Day 29, and Day 71.
Time Frame: Day 1, before dosing (baseline), and Day 29 and Day 71, after dosing.
Population: The Biological Activity Set (BAS) consisted of all FAS subjects who had at least 1 post-baseline skin biopsy (Visit 7, Visit 13), and received 2 doses of study drug. The primary analyses on biomarkers of disease activity obtained from biopsy were based on the BAS. Subjects were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 29 | 11
micrometer
  Baseline | 140.56 (57.623) | 124.95 (47.021)
  Change from Baseline in H&E Thickness to Day 29 | -14.90 (57.787) | -3.02 (51.589)
  Change from Baseline in H&E Thickness to Day 71 | -26.51 (88.676) | -6.01 (39.402)

3. Primary Outcome: Change From Baseline in Ratio of Active Atopic Dermatitis Messenger Ribonucleic Acid (mRNA) Expression (Normalized to Human Acidic Ribosomal Protein [hARP]) in Lesional Skin Biopsies
Description: Ratio of post-baseline/baseline value of messenger ribonucleic acid (mRNA) expression in lesional skin biopsies is reported.
Time Frame: 71 days
Population: The Biological Activity Set (BAS) consisted of all FAS participants who had at least 1 post-baseline skin biopsy (Visit 7, Visit 13), and received 2 doses of drug. The primary analyses on biomarkers of disease activity obtained from biopsy were based on the BAS. Participants were analyzed according to the treatment to which they were randomized.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 29 | 11
ratio
  CCL11/hARP | 0.67 [0.40 to 1.13] | 1.20 [0.5 to 2.9]
  CCL17/hARP | 0.62 [0.38 to 1.01] | 0.75 [0.34 to 1.67]
  CCL18/hARP | 0.75 [0.59 to 0.96] | 0.64 [0.43 to 0.96]
  CCL26/hARP | 0.81 [0.63 to 1.03] | 0.67 [0.45 to 1.01]
  CXCL10/hARP | 0.53 [0.36 to 0.79] | 0.85 [0.45 to 1.63]
  FOXP3/hARP | 0.88 [0.77 to 1.02] | 0.93 [0.74 to 1.16]
  INFg/hARP | 0.77 [0.48 to 1.23] | 1.34 [0.62 to 2.91]
  IL-23p40/hARP | 0.74 [0.52 to 1.04] | 0.71 [0.41 to 1.23]
  IL-5/hARP | 0.72 [0.39 to 1.32] | 0.67 [0.25 to 1.84]
  IL13/hARP | 0.96 [0.52 to 1.76] | 0.43 [0.16 to 1.11]
  IL17A/hARP | 1.01 [0.55 to 1.87] | 0.70 [0.25 to 1.96]
  IL22/hARP | 0.64 [0.42 to 0.99] | 0.47 [0.23 to 0.97]
  IL23p19/hARP | 0.92 [0.82 to 1.03] | 0.97 [0.81 to 1.17]
  K16/hARP | 0.58 [0.39 to 0.86] | 0.72 [0.37 to 1.38]
  MMP12/hARP | 0.58 [0.36 to 0.92] | 0.40 [0.19 to 0.85]
  OX40L/hARP | 1.04 [0.88 to 1.22] | 1.24 [0.97 to 1.58]
  S100A12/hARP | 0.42 [0.25 to 0.72] | 0.58 [0.24 to 1.39]
  S100A9/hARP | 0.51 [0.33 to 0.78] | 0.63 [0.31 to 1.28]
  TSLRP/hARP | 0.91 [0.79 to 1.05] | 0.84 [0.67 to 1.06]

4. Secondary Outcome: Percent Change in Eczema Area and Severity Index (EASI) Clinical Scores From Baseline
Description: In EASI, four disease characteristics of atopic dermatitis (erythema, edema/papulation, excoriation, and lichenification) are assessed for severity on a scale of 0 (absent), 1 (mild), 2 (moderate), 3 (severe). The scores are added up for each of the four body regions (Head and neck, trunk, arms, and legs). The assigned percentages of body surface area (BSA) for each section of the body are 10% for head and neck, 20% for arms, 30% for trunk, and 40% for legs, respectively. Each subtotal score is multiplied by the BSA represented by that region. In addition, an area score of 0 to 6 is assigned for each body region, depending on the percentage of AD-affected skin in that area: 0 (none), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Each of the body area scores are multiplied by the area affected. The resulting EASI score ranges from 0 to 72 points, with the highest score indicating worse severity of AD.
Time Frame: Day 4, Day 29, Day 57, Day 71
Population: Full Analysis Set (FAS): The FAS consisted of all participants who were randomized and received at least 1 partial or full dose of study treatment. The FAS population was used for the analysis of the efficacy data not obtained from skin biopsy. Participants were analyzed according to the treatment by which they were randomized.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 46 | 16
percentage of change from baseline
  Percent Change from Baseline to Visit 3 (Day 4) | -9.80 (14.253) | -11.33 (16.835)
  Percent Change from Baseline to Visit 7 (day 29) | -38.72 (36.148) | -32.40 (31.918)
  Percent Change from Baseline to Visit 12 (day 57) | -61.00 (31.951) | -39.54 (46.791)
  Percent Change from Baseline to Visit 13 (day 71) | -67.35 (23.107) | -38.22 (37.865)

5. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Clinical Score of 0 or 1
Description: The IGA is an assessment scale used in clinical studies to determine severity of AD based on a 5-point scale ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 4, Day 29, Day 57, Day 71
Population: N is the number of participants in the respective treatment group. Numbers and percentages calculated at each visit are based on the number of participants achieving IGA score of 0 or 1 among those evaluable participants at each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 46 | 16
Participants
  Visit 3 (day 4): number analyzed (Participants) | 0 | 0
  Visit 3 (day 4) | 0 | 0
  Visit 7 (day 29): number analyzed (Participants) | 34 | 0
  Visit 7 (day 29) | 2 | 0
  Visit 12 (day 57): number analyzed (Participants) | 25 | 10
  Visit 12 (day 57) | 6 | 2
  Visit 13 (day 71): number analyzed (Participants) | 23 | 8
  Visit 13 (day 71) | 6 | 1

6. Secondary Outcome: Pharmacokinetics of GBR 830 in Terms of Cmax After First and Second Dose.
Description: Pharmacokinetics in terms of Cmax (maximum observed concentration after second [last] dosing interval) was estimated after the first and second dose.
Time Frame: Blood samples were collected on Day 1 and Day 29: pre-dose (15 mins), end of infusion (1 hour) and 1.5, 2, 72, and 504 hours post start of infusion
Population: The Pharmacokinetic Analysis Set (PKAS) consisted of the subset of the Safety Analysis Set population for which sufficient serum concentration data were available to facilitate derivation of at least 1 PK parameter, and the time (HH:MM) of dosing on the day of sampling was known for at least 1 of the dosing visits.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | GBR 830
Number analyzed (Participants) | 45
microgram/mL
  Cmax after First Dose | 303 (29)
  Cmax after Second Dose | 352 (29)

7. Secondary Outcome: Pharmacokinetics of GBR 830 in Terms of AUC0-tau After the First and Second Dose.
Description: Pharmacokinetics in terms of AUC0-tau [Trapezoid calculation of area under the serum drug concentration-time curve from time zero (pre dose time point of the infusion) to the end of the dosing interval] was estimated.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/mL
Arm/Group | GBR 830
Number analyzed (Participants) | 40
microgram*hour/mL
  AUC0-tau after the First Dose | 57217 (26)
  AUC0-tau after the Second Dose | 69670 (29)

8. Secondary Outcome: Number of Participants Positive or Negative for Anti-drug Antibodies (ADA) to GBR 830 to Evaluate Immunogenicity
Description: Blood samples were collected at time points to detect anti-drug antibodies (ADAs) to GBR 830, as per procedures similar to collection of PK samples. Antibodies of GBR 830 were detected and confirmed using a validated enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Samples collected for immunogenicity analysis at Baseline (pre-dose), and at Day 15, Day 29 (pre-dose), Day 57, and Day 85.
Population: The Safety Analysis Set consisted of all particpants who took at least 1 full or partial dose of study treatment and were used in the assessment and reporting of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | GBR 830 | Placebo
Number analyzed (Participants) | 46 | 16
Participants
  Positive | 6 | 1
  Negative | 40 | 15

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of signing the informed consent form (ICF) until the follow up for a total duration of 16 weeks.
Description: A total of 64 eligible participants were randomized to receive either GBR 830 or corresponding placebo. Two participants assigned to GBR 830 withdrew informed consent before dosing. Therefore, a total of 62 subjects were included in the Full Analysis Set and Safety Analysis Set.
Arm/Group | GBR 830 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/16
Other Adverse Events (participants affected / at risk) | 21/46 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBR 830 (N=46) | Placebo (N=16)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBR 830 (N=46) | Placebo (N=16)
Nasopharyngitis (Infections and infestations) | 4 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2)
post procedural infection (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 4 (5)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 2 (4) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT02683928/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT02683928/SAP_001.pdf